CLINICAL TRIAL: NCT01574326
Title: A 2-Week, Randomized, Placebo-Controlled, Fixed Dose Period Followed by a 6-Month, Single-Arm, Open-Label, Dose Titration Period Study to Investigate the Efficacy and Safety of Sevelamer Carbonate in Hyperphosphatemic Pediatric Patients With Chronic Kidney Disease
Brief Title: An Efficacy and Safety Study of Sevelamer Carbonate in Hyperphosphatemic Pediatric Participants With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SVCARB07609; 2011-002329-23 (EudraCT Number); DRI12793 (Other: Genzyme Corporation)
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Hyperphosphatemia; Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Pediatric; Sevelamer Carbonate; Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia; Renal Insufficiency, Chronic | interventions — Sevelamer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FDP-Placebo for Sevelamer Carbonate, DTP-Sevelamer Carbonate (Placebo Comparator): Participants received placebo for 2 weeks during the fixed dose period (FDP). Participants received sevelamer carbonate for 26 weeks in dose titration period (DTP).
  Interventions: Drug: Placebo; Drug: Sevelamer carbonate
- FDP-Sevelamer Carbonate, DTP-Sevelamer Carbonate (Experimental): Participants received sevelamer carbonate for 2 weeks during the FDP of the study. Participants received sevelamer carbonate for an additional 26 weeks in DTP.
  Interventions: Drug: Placebo; Drug: Sevelamer carbonate

INTERVENTIONS:
Drug: Placebo — Placebo for 0.8 g sachets of powder for oral suspension or 800 mg tablets
Drug: Sevelamer carbonate — 0.8 g sachets of powder for oral suspension or 800 mg tablets
  Other Names: Renvela®

SUMMARY:
Objective: In hyperphosphatemic pediatric participants with chronic kidney disease (CKD) to

* Evaluate the safety and tolerability of sevelamer carbonate
* Evaluate the efficacy of sevelamer carbonate on the control of serum phosphorus

DETAILED DESCRIPTION:
The study was divided into 3 periods: a phosphate binder washout Period; a randomized, double-blind, placebo-controlled, Fixed Dose Period; and an open-label, sevelamer carbonate Dose Titration Period.

ELIGIBILITY:
Inclusion Criteria:

* The participant had CKD requiring dialysis or CKD not on dialysis with an estimated glomerular filtration rate (GFR) <60 mL/min/1.73 m^2 based on central laboratory results.
* The participant had a serum phosphorus level greater than the age appropriate upper limit of normal based on central laboratory results.

Exclusion Criteria:

* The participant had active dysphagia, swallowing disorders or a predisposition to or current bowel obstruction, ileus or severe gastrointestinal motility disorder(s) including severe constipation, or major gastrointestinal tract surgery.
* The participant had a non-renal case of hyperphosphatemia.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2012-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (32):
- United States (23):
  - Investigational Site Number 8003, Birmingham, Alabama
  - Investigational Site Number 8005, Birmingham, Alabama
  - Investigational Site Number 8013, Los Angeles, California
  - Investigational Site Number 8014, San Francisco, California
  - Investigational Site Number 8025, Orlando, Florida
  - Investigational Site Number 8007, Atlanta, Georgia
  - Investigational Site Number 8019, Iowa City, Iowa
  - Investigational Site Number 8012, Baltimore, Maryland
  - Investigational Site Number 8008, Boston, Massachusetts
  - Investigational Site Number 8020, Detroit, Michigan
  - Investigational Site Number 8022, Kansas City, Missouri
  - Investigational Site Number 8023, St Louis, Missouri
  - Investigational Site Number 8017, Livingston, New Jersey
  - Investigational Site Number 8018, Buffalo, New York
  - Investigational Site Number 8009, Greenville, North Carolina
  - Investigational Site Number 8010, Portland, Oregon
  - Investigational Site Number 8011, Philadelphia, Pennsylvania
  - Investigational Site Number 8026, Dallas, Texas
  - Investigational Site Number 8016, Houston, Texas
  - Investigational Site Number 8001, San Antonio, Texas
  - Investigational Site Number 8002, Charlottesville, Virginia
  - Investigational Site Number 8027, Richmond, Virginia
  - Investigational Site Number 8006, Seattle, Washington
- France (3):
  - Investigational Site Number 8101, Bordeaux
  - Investigational Site Number 8102, Bron
  - Investigational Site Number 8103, Paris
- Germany (2):
  - Investigational Site Number 8201, Berlin
  - Investigational Site Number 8202, Marburg
- Lithuania (2):
  - Investigational Site Number 8302, Kaunas
  - Investigational Site Number 8301, Vilnius
- Poland (2):
  - Investigational Site Number 8402, Gdansk
  - Investigational Site Number 8401, Krakow

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 29 centers in 4 countries. A total of 128 participants were screened between 11 May 2012 and 14 November 2014. Of whom, 101 participants were randomized and 27 were screen failures.
Pre-assignment Details: Participants were stratified in (1:1) by screening body surface area (BSA) (≥1.2 vs <1.2 m^2) & qualifying serum phosphorus (≥7.0 vs <7.0 mg/dL) to get sevelamer carbonate or placebo in 2 week fixed dose period (FDP). Following FDP, participants entered 26-week dose titration period (DTP) during which all participants received sevelamer carbonate.
Groups:
- FDP-Placebo for Sevelamer Carbonate, DTP-Sevelamer Carbonate: Participants received placebo for sevelamer carbonate for 2 weeks in FDP and sevelamer carbonate for 26 weeks in DTP. Placebo matched to sevelamer carbonate 3 times a day (TID) for 2 weeks in FDP: 0.4 g TID for BSA <0.75 m^2 or 0.8 g TID for BSA ≥0.75 to < 1.2 m^2 as powder for oral suspension (POS) & 1.6 g TID for BSA ≥1.2 m^2 as POS/tablets as per participant's preference. If a child ate <3 meals/snacks per day, dose was given with meals/snacks. In DTP, starting dose of sevelamer carbonate was based on screening BSA & same as prescribed during FDP. Dose was titrated up/down every 2 weeks for 6 weeks & then every 4 weeks to achieve a serum phosphorus level within age appropriate normal values or up to maximum dose as per Investigator's opinion. Dose titrations were based on BSA category: 0.2 g TID for BSA <0.75 m^2, 0.4 g TID for BSA ≥0.75 to < 1.2 m^2 & 0.8 g TID for BSA ≥1.2 m^2 (smaller titrations were permitted but could not be <0.2 g TID with meals/snacks).
- FDP-Sevelamer Carbonate, DTP-Sevelamer Carbonate: Participants received sevelamer carbonate 0.4 g TID or 0.8 g TID or 1.6 g TID (based on screening BSA category) for 2 weeks in FDP and then continued to receive sevelamer carbonate in DTP. Sevelamer carbonate for 2 weeks in FDP: 0.4 g TID for BSA <0.75 m^2 or 0.8 g TID for BSA ≥0.75 to < 1.2 m^2 as POS or 1.6 g TID for BSA ≥1.2 m^2 either as POS or tablets as per participant's preference. If a child ate <3 meals/snacks per day, dose was given with meals/snacks. In DTP, starting dose of sevelamer carbonate was based on screening BSA & same as dose prescribed during FDP. Dose was titrated up/down every 2 weeks for 6 weeks & then every 4 weeks to achieve a serum phosphorus level within age appropriate normal values or up to maximum dose as per Investigator's opinion. Dose titrations were based on BSA category: by 0.2 g TID for BSA <0.75 m^2, 0.4 g TID for BSA ≥0.75 to <1.2 m^2 & 0.8 g TID for BSA ≥1.2 m^2 (smaller titrations were permitted but could not be <0.2 g TID with meal/snacks).
Period: Overall Study
Arm/Group | FDP-Placebo for Sevelamer Carbonate, DTP-Sevelamer Carbonate | FDP-Sevelamer Carbonate, DTP-Sevelamer Carbonate
Started | 51 | 50
Treated | 51 | 49
Completed | 35 | 31
Not Completed | 16 | 19
Not completed — Randomized but not treated | 0 | 1
Not completed — Withdrawal by Participant | 2 | 4
Not completed — Physician Decision | 5 | 3
Not completed — Adverse Event | 1 | 3
Not completed — Other: Mainly kidney transplant | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- FDP-Placebo for Sevelamer Carbonate, DTP-Sevelamer Carbonate: Participants received placebo for sevelamer carbonate for 2 weeks in FDP and sevelamer carbonate for 26 weeks in DTP. Placebo matched to sevelamer carbonate TID for 2 weeks in FDP: 0.4 g TID for BSA <0.75 m^2 or 0.8 g TID for BSA ≥0.75 to < 1.2 m^2 POS and 1.6 g TID for BSA ≥1.2 m^2 as POS/tablets as per participant's preference. If a child ate <3 meals/snacks per day, dose was given with meals/snacks. In DTP, starting dose of sevelamer carbonate was based on screening BSA & same as prescribed during FDP. Dose was titrated up/down every 2 weeks for 6 weeks & then every 4 weeks to achieve a serum phosphorus level within age appropriate normal values or up to maximum dose as per Investigator's opinion. Dose titrations were based on BSA category: 0.2 g TID for BSA <0.75 m^2, 0.4 g TID for BSA ≥0.75 to < 1.2 m^2 & 0.8 g TID for BSA ≥1.2 m^2 (smaller titrations were permitted but could not be <0.2 g TID with meals/snacks).
- Total: Total of all reporting groups
Arm/Group | FDP-Placebo for Sevelamer Carbonate, DTP-Sevelamer Carbonate | FDP-Sevelamer Carbonate, DTP-Sevelamer Carbonate | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] — Age continuous is reported here for safety set: N= 51 and N=49 for 'FDP-Placebo for sevelamer carbonate, DTP-Sevelamer carbonate' and 'FDP-Sevelamer carbonate, DTP-Sevelamer carbonate' arms respectively. All enrolled participants who were treated with at least 1 dose of study drug were included in the safety set.
  years | 14.3 (3.11) | 13.9 (2.75) | 14.1 (2.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 33 | 31 | 64

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Week 0) to Week 2 in Serum Phosphorus
Description: Full analysis set for fixed dose period (FAS-FDP) participants were analyzed according to their randomized treatment. The change in serum phosphorus (mg/dL) from baseline to week 2 was calculated.
Time Frame: Baseline, Week 2
Population: FAS-FDP population included all treated participants with a baseline phosphorus value and at least 1 post-baseline assessment after the first dose of study drug and on or before Week 2. Three participants (1 in sevelamer carbonate group and 2 in placebo group) were excluded from FAS-FDP due to no baseline phosphorus value at week 2.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- FDP-Placebo for Sevelamer Carbonate: Participants received placebo for sevelamer carbonate for first 2 weeks in FDP.
- FDP-Sevelamer Carbonate: Participants received sevelamer carbonate 0.4 g TID or 0.8 g TID or 1.6 g TID (based on the screening BSA category) for 2 weeks in FDP.
Arm/Group | FDP-Placebo for Sevelamer Carbonate | FDP-Sevelamer Carbonate
Number analyzed (Participants) | 49 | 48
mg/dL
  At Baseline | 7.2 (1.841) | 7.2 (2.09)
  At Week 2 | 7.24 (2.029) | 6.34 (1.306)
  Change from baseline to Week 2 | 0.04 (1.478) | -0.87 (1.649)
Statistical Analysis 1: Comparison: FDP-Placebo for Sevelamer Carbonate vs FDP-Sevelamer Carbonate; Primary efficacy endpoint, change from baseline to Week 2 in serum phosphorus, was compared between treatment groups using analysis of covariance (ANCOVA) with baseline phosphorus and screening BSA as covariates and fixed effect for treatment. No center effect was included in the model. The estimate of the treatment difference (Sevelamer Carbonate - Placebo) and its 95% CI were presented. Significance was to be declared if the p-value was ≤0.05; Test type: Superiority or Other; p = 0.001, ANCOVA; Threshold for significance ≤ 0.05; Least square (LS) mean difference = -0.9, 95% CI 2-sided [-1.44 to -0.37]

2. Primary Outcome: Treatment - Emergent Adverse Events (AEs)
Description: A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect. AEs from the time of signing the informed consent through the end of the study for all participants. SAEs occurring during the 15 days following study completion or early termination were also to be collected.
Time Frame: Up to 32 weeks (up to 4 weeks washout period, 2 weeks FDP and 26 weeks DTP)
Population: Analysis was performed on safety set, which included all enrolled participants who received at least 1 dose of study drug. Participants were analyzed according to actual received treatment.
Measure: Number; unit: participants
Groups:
- FDP- Placebo for Sevelamer Carbonate; DTP- Sevelamer Carbonate: Participants received placebo for sevelamer carbonate for first 2 weeks in FDP. Thereafter, participants received sevelamer carbonate for 26 weeks in DTP.
- FDP-Sevelamer Carbonate, DTP-Sevelamer Carbonate: Participants received sevelamer carbonate 0.4 g TID or 0.8 g TID or 1.6 g TID (based on the screening BSA category) for 2 weeks in FDP. Thereafter, participants continued to receive sevelamer carbonate for 26 weeks in DTP based on the screening BSA category.
Arm/Group | FDP- Placebo for Sevelamer Carbonate; DTP- Sevelamer Carbonate | FDP-Sevelamer Carbonate, DTP-Sevelamer Carbonate
Number analyzed (Participants) | 51 | 49
participants
  Any AE: FDP | 20 | 19
  AE related: FDP | 3 | 2
  Any SAE: FDP | 1 | 4
  SAE related: FDP | 0 | 0
  Any AE Leading to Study Drug Discontinuation: FDP | 1 | 1
  Any AE: DTP | 42 | 35
  AE related: DTP | 9 | 4
  Any SAE: DTP | 14 | 17
  SAE related: DTP | 2 | 2
  Any AE Leading to Study Drug Discontinuation: DTP | 0 | 3
  Deaths | 0 | 0

3. Secondary Outcome: Change From Baseline (Week 0) to Week 28/Early Termination in Serum Phosphorus
Description: Full analysis set for dose titration period (FAS-DTP) participants were analyzed according to their randomized treatment. The change in serum phosphorus (mg/dL) from baseline to Week 28/Early Termination was calculated.
Time Frame: Baseline, Week 28/Early Termination
Population: FAS-DTP population included all treated participants with a baseline phosphorus value and at least 1 post-baseline phosphorus assessment after Week 2. Five participants (3 in sevelamer carbonate group and 2 in the placebo group) were excluded from the FAS-DTP due to no baseline phosphorus value or no phosphorus assessment after Week 2.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- FDP- Placebo for Sevelamer Carbonate; DTP- Sevelamer Carbonate: Participants received placebo for sevelamer carbonate for first 2 weeks in FDP. Thereafter participants received sevelamer carbonate for 26 weeks in DTP.
- FDP-Sevelamer Carbonate, DTP-Sevelamer Carbonate: Participants received sevelamer carbonate 0.4 g TID or 0.8 g TID or 1.6 g TID (based on the screening BSA category) for 2 weeks in FDP. Thereafter, participants continued to receive sevelamer carbonate for 26 weeks in DTP.
Arm/Group | FDP- Placebo for Sevelamer Carbonate; DTP- Sevelamer Carbonate | FDP-Sevelamer Carbonate, DTP-Sevelamer Carbonate
Number analyzed (Participants) | 49 | 46
mg/dL
  At Baseline (Week 0) | 7.05 (1.797) | 7.28 (2.103)
  At Week 28 / Early Termination | 5.92 (1.612) | 6.04 (1.878)
  Change from Baseline to Week 28/Early Termination | -1.13 (2.061) | -1.23 (2.206)

ADVERSE EVENTS:
Time Frame: All AEs were collected from signature of informed consent form up to final visit regardless of seriousness or relationship to investigational product. SAEs occurring during 15 days following study completion or early termination were also to be collected.
Description: Reported AEs are treatment emergent adverse events (includes non-serious AEs and SAEs as applicable) that is AE that developed/worsened during the 'on treatment period' (from the first dose of study drug up to end of study period). Analysis was performed on safety set.
Groups:
- FDP - Placebo: Participants exposed to placebo (for sevelamer carbonate) for first 2 weeks in FDP (median exposure of 15 days).
- FDP - Sevelamer Carbonate: Participants exposed to sevelamer carbonate 0.4 g TID or 0.8 g TID or 1.6 g TID (based on the screening BSA category) for first 2 weeks in FDP (median exposure of 15 days).
- DTP - Sevelamer Carbonate: Participants who received placebo and participants who received sevelamer carbonate in FDP received sevelamer carbonate for 26 weeks in DTP (median exposure of 183.5 days in participants who were on sevelamer carbonate in FDP and 183 days in participants who were on placebo in FDP).
Arm/Group | FDP - Placebo | FDP - Sevelamer Carbonate | DTP - Sevelamer Carbonate
Serious Adverse Events (participants affected / at risk) | 1/51 | 4/49 | 31/100
Other Adverse Events (participants affected / at risk) | 6/51 | 7/49 | 57/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FDP - Placebo (N=51) | FDP - Sevelamer Carbonate (N=49) | DTP - Sevelamer Carbonate (N=100)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Device dislocation (General disorders) | 0 | 0 | 1
Device malfunction (General disorders) | 0 | 0 | 2
Device occlusion (General disorders) | 0 | 1 | 1
Extravasation (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 3
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 | 0 | 1
Kidney transplant rejection (Immune system disorders) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 2
Catheter site infection (Infections and infestations) | 0 | 0 | 1
Fungal peritonitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 2
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Urosepsis (Infections and infestations) | 0 | 0 | 1
Vaginitis chlamydial (Infections and infestations) | 0 | 0 | 1
Varicella zoster virus infection (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural constipation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 | 0 | 1
Oliguria (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 2 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FDP - Placebo (N=51) | FDP - Sevelamer Carbonate (N=49) | DTP - Sevelamer Carbonate (N=100)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 13
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 9
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 8
Nausea (Gastrointestinal disorders) | 2 | 0 | 15
Vomiting (Gastrointestinal disorders) | 3 | 0 | 19
Catheter site pain (General disorders) | 0 | 0 | 6
Pyrexia (General disorders) | 0 | 1 | 16
Seasonal allergy (Immune system disorders) | 0 | 0 | 6
Nasopharyngitis (Infections and infestations) | 0 | 0 | 6
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 8
Dizziness (Nervous system disorders) | 0 | 1 | 7
Headache (Nervous system disorders) | 2 | 2 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 7
Hypertension (Vascular disorders) | 0 | 1 | 7
Hypotension (Vascular disorders) | 1 | 0 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.